CLINICAL TRIAL: NCT02624635
Title: Effects of Adding Hip Strengthening to Manual Therapy for Heel Pain Patients
Brief Title: Hip Strengthening and Manual Therapy for Heel Pain Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of the lack of personnel and the recruitment failure of participants.
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1174-3946
Record Dates: First submitted 2015-12-01; First posted 2015-12-08 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Plantar Fasciitis
Keywords: Manual Therapy; Pain; Hip; Muscle Strength
MeSH Terms: conditions — Fasciitis, Plantar; Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manual Therapy (Active Comparator): The treatment for this group will be manual therapy.
  Interventions: Other: Manual Therapy
- Manual Therapy and Hip Strengthening (Experimental): It will be done the same treatment performed in group 1 plus the strengthening of the muscles of the hip.
  Interventions: Other: Manual Therapy and Hip Strengthening

INTERVENTIONS:
Other: Manual Therapy — The scheme established for that intervention is as follows: joint manipulation passive ankle and foot, myofascial release technique (gastrocnemius, soleus muscle and plantar fascia), neural mobilization (nerve tibial) and stretching the plantar region and sural triceps, following the recommendations described by Mcpoil et al. (2008).
  Arms: Manual Therapy
Other: Manual Therapy and Hip Strengthening — It will be done the same treatment performed in group 1 plus the strengthening of the muscles of the hip (iliac muscle, psoas, gluteus maximus, gluteus medius and gluteus minimus) and the treatment schedule established for this intervention is the use of exercises with progressive resistance. Will be performed 3 sets of 10 reps with 30 seconds rest between each set, according to the guidelines of the American College of Sports Medicine (ACSM, 2014). The home exercises consist of repeating the same procedures performed for supervised strengthening. The calculation of the ideal individual load will be carried by Brzycki formula, i.e. one repetition maximum (1RM) = weight ÷ [1.0278 - (0.0278 x number of repetitions)] as was used by (Shirazi et al., 2007).
  Arms: Manual Therapy and Hip Strengthening

SUMMARY:
The purpose of this study is to compare the effects of manual therapy and of manual therapy associated with hip strengthening in the recovery of patients with heel pain.

Heel pain decreases function, balance, walking and can cause change in the movement pattern. This alterations can induce a deficit in motor control of other structures as knee and hip. There is an importance to compare the effects of manual therapy and manual therapy associated with hip strengthening on the recover of patients with heel pain.

DETAILED DESCRIPTION:
After the initial assessment and data collection, participants will be randomly assigned to one of two intervention groups. Randomization will be held electronically in http://graphpad.com/quickcalcs/index.cfm site by simple random sampling. Patients will be treated for a maximum of 10 sessions, each session lasting about 40 minutes and each week two sessions. The maximum duration of treatment is 3 months. A physical therapist will be responsible for the screening of eligible patients and the random allocation of participants A second professional will be responsible for physical therapy initial and final evaluation and will be blind to the interventions. A third physical therapist will perform the interventions. The physiotherapist in charge of intervention will be blind to the initial and final evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heel pain, that increases on the first steps after a period without activity and with long periods on standing position, regardless of age and gender and that didn't went under any physiotherapeutic treatment in the last 3 months.

Exclusion Criteria:

* Patients who have a history of surgery on the lower limb on the past 6 months; patients with bilateral heel pain; patients under psychiatric treatment; patients that went under a manual therapy scheme treatment for heel pain before; rheumatic syndromes; patients who receive some benefit labor or patients underage.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Level of intensity of pain | Up to three months
  Level of intensity of pain assessed through the numerical pain scale.

SECONDARY OUTCOMES:
Functional Status | Up to three months
  Level of disability of the lower limb assessed through Lower Extremity Functional Scale.
Pressure pain threshold | Up to three months
  Pressure pain threshold assessed through the algometer.

CONTACTS AND LOCATIONS:
Overall Officials: Leandro AC Nogueira, PhD, Principal Investigator — Centro Universitário Augusto Motta
Locations (1):
- Hospital Universitário Gaffréé Guinle, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Acevedo JI, Beskin JL. Complications of plantar fascia rupture associated with corticosteroid injection. Foot Ankle Int. 1998 Feb;19(2):91-7. doi: 10.1177/107110079801900207. PMID 9498581
- [Background] Ajimsha MS, Binsu D, Chithra S. Effectiveness of myofascial release in the management of plantar heel pain: a randomized controlled trial. Foot (Edinb). 2014 Jun;24(2):66-71. doi: 10.1016/j.foot.2014.03.005. Epub 2014 Mar 21. PMID 24703512
- [Background] Moore AR, Eccleston C, Derry S, Wiffen P, Bell RF, Straube S, McQuay H; ACTINPAIN writing group of the IASP Special Interest Group (SIG) on Systematic Reviews in Pain Relief and the Cochrane Pain, Palliative and Supportive Care Systematic Review Group editors. "Evidence" in chronic pain--establishing best practice in the reporting of systematic reviews. Pain. 2010 Sep;150(3):386-389. doi: 10.1016/j.pain.2010.05.011. Epub 2010 Jun 2. No abstract available. PMID 20627575
- [Background] Babcock MS, Foster L, Pasquina P, Jabbari B. Treatment of pain attributed to plantar fasciitis with botulinum toxin a: a short-term, randomized, placebo-controlled, double-blind study. Am J Phys Med Rehabil. 2005 Sep;84(9):649-54. doi: 10.1097/01.phm.0000176339.73591.d7. PMID 16141740
- [Background] Bergmann JN. History and mechanical control of heel spur pain. Clin Podiatr Med Surg. 1990 Apr;7(2):243-59. PMID 2189536
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Buch M, Knorr U, Fleming L, Theodore G, Amendola A, Bachmann C, Zingas C, Siebert WE. [Extracorporeal shockwave therapy in symptomatic heel spurs. An overview]. Orthopade. 2002 Jul;31(7):637-44. doi: 10.1007/s00132-002-0323-z. German. PMID 12219661